CLINICAL TRIAL: NCT01061580
Title: Dose Response Study of Autologous Concentrated Bone Marrow Nucleated Cell Therapy for Congestive Heart Failure Patients Undergoing Treatment With Coronary Artery Bypass Grafting (CABG) Surgery
Brief Title: BMAC Enhanced Coronary Artery Bypass Grafting (CABG)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Harvest Technologies (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2009-1
Record Dates: First submitted 2009-12-16; First posted 2010-02-03 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Congestive Heart Failure
Keywords: Bone Marrow Concentrate; CABG; Cardiac; Stem Cell
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CABG plus BMAC Injection (Experimental): Injection of Bone Marrow Aspirate Concentrate (BMAC) into ischemic myocardium following CABG during the same open procedure
  Interventions: Device: Harvest SmartPReP2 BMAC System

INTERVENTIONS:
Device: Harvest SmartPReP2 BMAC System — Injection of 10, 15, or 20 cc of BMAC

SUMMARY:
Injection of concentrated bone marrow cells into the myocardium during CABG procedure.

DETAILED DESCRIPTION:
Injection of autologous concentrated bone marrow cells into the myocardium during CABG procedure.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to be enrolled in the trial:

* Age 18 years and ability to understand the planned treatment.
* Patients with ischemic congestive heart failure requiring by pass surgery
* Congestive heart failure with ejection fraction 40%.
* Serum bilirubin, SGOT and SGPT 2.5 time the upper level of normal.
* Serum creatinine < 3.0 or no dialysis.
* NYHA performance status > 3.
* Negative pregnancy test (in women with childbearing potential).
* Subject has read and signed the IRB approved Informed Consent form
* Hematocrit ≥ 28.0%, White Blood Cell count ≤ 14,000, Platelet count ≥ 50,000, Creatinine ≤ 3.0 mg / Dl, and/or no dialysis, INR ≤ 1.6 unless on Coumadin, or PTT <1.5 x control (to avoid bleeding complications) Patients on Coumadin will be corrected prior to the procedure and must have an INR<1.6 at the time of randomization/surgery

Exclusion Criteria:

Subjects will be excluded if they meet any of the exclusion criteria:

* Female who is pregnant or nursing, or of child bearing potential and is not using a reliable birth control method, or who intend to become pregnant during the tenure of this study.
* History of Prior Radiation Exposure for oncological treatment.
* History of Bone Marrow Disorder (especially NHL, MDS) that prohibit transplantation.
* History of abnormal Bleeding or Clotting.
* History of Liver Cirrhosis.
* Acute Myocardial Infarction < 4 weeks from treatment date.
* Known active malignancy or results outside of normal limits from the following tests: PAP, Chest X-ray, PSA, Mammogram, Hemocult unless follow-up studies reveal patient to be cancer free.
* Active clinical infection being treated by antibiotics within one week of enrollment
* Terminal renal failure with existing dependence on dialysis
* Inability or unwillingness to comply with the treatment protocol, follow-up, research tests, or give consent.
* Unable to have 250cc bone marrow harvested.
* Medical risk that precludes anesthesia or ASA Class 5
* History of ventricular arrhythmia if AICD is not present.
* History of ventricular aneurysm.
* Concurrent surgery such as CABG with valve surgery.
* Minimally Invasive bypass surgery
* Life expectancy <6 months due to concomitant illnesses
* Treatment with immunosuppressant drugs (including Prednisone > 5 mg per day)
* Patients undergoing urgent by pass surgical procedure
* Patients with HGB A1C > 8.5%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-05; Primary Completion 2012-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Changes in left ventricular function | 12 months

SECONDARY OUTCOMES:
QOL (Rand 36; Minnesota Living with Heart Failure Questionnaire) | 12 months
NYHA or CCS classification evaluation | 12 months
Changes in left ventricular ejection fraction | 12 months
Changes in left ventricular end-diastolic volume | 12 months
Safety | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Naresh Trehan, MD, Principal Investigator — Medanta-The Medicity
Locations (1):
- Medanta The Medicity, Gurgaon, Haryana, India